CLINICAL TRIAL: NCT01822366
Title: Improving Health Outcomes by Preventing HIV/STD Risk
Brief Title: Randomized Controlled Trial of Trauma-focused CBT in Tanzania and Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Tanzania Women Research Foundation (TAWREF) (Unknown); Ace Africa (Other); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00039770; R01MH096633 (NIH)
Record Dates: First submitted 2013-03-25; First posted 2013-04-02 (Estimated); Results first posted 2019-05-23 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Childhood Traumatic Grief; Post Traumatic Stress; Post Traumatic Stress Disorder; Depressive Symptoms; Behavioral Problems; Child Overall Daily Functioning; Child and Guardian Relationship
Keywords: Children; Adolescents; Trauma-focused Cognitive Behavioral Therapy (TF-CBT); Low- and Middle-Income Countries (LMIC); Randomized Controlled Trial (RCT); Evidence-Based Practice (EBP); Childhood Traumatic Grief (CTG); Post-Traumatic Stress Disorder (PTSD); Kenya; Tanzania; East Africa; Mental Health
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Problem Behavior; Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care Comparison Condition (No Intervention): Half of the participating children/guardian dyads will receive no intervention (usual care) to serve as a control.
- Trauma-focused CBT group therapy (Experimental): Half of the participating children/guardian dyads will receive the 12-week Trauma-focused Cognitive Behavioral Therapy (TF-CBT) group treatment.
  Interventions: Behavioral: Trauma-focused Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Trauma-focused Cognitive Behavioral Therapy
  Arms: Trauma-focused CBT group therapy

SUMMARY:
The primary goal is to study the effectiveness of Trauma-focused Cognitive Behavioral Therapy (TF-CBT) in treating traumatic grief and traumatic stress for orphaned children and young adolescents in two East African sites with high prevalence HIV, Moshi, Tanzania (TZ) and Bungoma, Kenya (KE), through a randomized controlled trial (RCT). In a previous feasibility study of TF-CBT with orphans in Tanzania, the investigators have found a group-based TF-CBT intervention to be feasible and acceptable, with promising clinical outcomes. In the feasibility study, lay counselors with no prior mental health experience delivered the intervention with training and supervision by our team of mental health and TF-CBT experts.

Building on this initial study, the investigators are conducting a RCT to test the effectiveness of TF-CBT for traumatic grief and traumatic stress compared to receipt of usual care orphan services in TZ and KE. The study involves collaboration with HIV/AIDS grassroots organizations and local Co-Investigators in TZ and KE, both of whom are longstanding collaborators with the investigators' US team and are located in mixed urban and rural areas, allowing examination of effectiveness in two countries and two settings (urban/rural). Using a task-shifting approach, in which lay individuals are trained as counselors, the investigators will train six counselors in each country, who deliver 20 groups in each site (8 rural, 12 urban), resulting in 320 children and adolescents (ages 7-13) who receive TF-CBT and 320 who receive usual care. Outcomes for children are assessed at 12-14 weeks (i.e., corresponding with the end of TF-CBT), 6-months post-treatment, and 12-months post-treatment. TF-CBT experts from the investigators' team partner with the lay counselors from the feasibility study (e.g., local trainers) to train the TZ and KE counselors, and these local trainers provide the TF-CBT supervision, while supervised themselves by the US-based TF-CBT and mental health experts. The investigators expect this trial to yield recommendations regarding an effective intervention for orphans that is acceptable, feasible, and includes local responsibility as a means to enhance potential sustainability in Low- and Middle-Income Countries (LMICs). Findings will inform other efforts to scale up mental health interventions to address the substantial mental health gap.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 7-13 living in Moshi, Tanzania or Bungoma, Kenya who have had one or both parents die since they were 3 years old or older.
* Children must have scores on study measures indicating they have symptoms of traumatic grief and/or traumatic stress.
* Children must be living with an adult guardian who is willing to participate in 12 weekly group sessions.
* Adult guardians of eligible children.

Exclusion Criteria:

* Living in an institution (not with a guardian).
* Parent(s) died before child was 3 years old.

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1280 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Dorsey, PhD, Principal Investigator — University of Washington; Kate Whetten, PhD, MPH, Principal Investigator — Duke University
Locations (3):
- University of Washington Department of Psychology, Seattle, Washington, United States
- Action in the Community Environment (ACE) Africa, Bungoma, Kenya
- Tanzania Women Research Foundation (TAWREF), Moshi, Tanzania

REFERENCES:
- [Derived] Dorsey S, Lucid L, Martin P, King KM, O'Donnell K, Murray LK, Wasonga AI, Itemba DK, Cohen JA, Manongi R, Whetten K. Effectiveness of Task-Shifted Trauma-Focused Cognitive Behavioral Therapy for Children Who Experienced Parental Death and Posttraumatic Stress in Kenya and Tanzania: A Randomized Clinical Trial. JAMA Psychiatry. 2020 May 1;77(5):464-473. doi: 10.1001/jamapsychiatry.2019.4475. PMID 31968059
- See also: Pamoja Tunaweza (Together We Can) — http://depts.washington.edu/risemh/pamoja-tunaweza-together-we-can/

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care Comparison Condition - Children; Usual Care Comparison Condition - Caregivers: Half of the participating children/guardian dyads will receive no intervention (usual care) to serve as a control.
- Trauma-focused CBT Group Therapy - Children; Trauma-focused CBT Group Therapy - Caregivers: Half of the participating children/guardian dyads will receive the 12-week Trauma-focused Cognitive Behavioral Therapy (TF-CBT) group treatment.
  Trauma-focused Cognitive Behavioral Therapy
Period: Overall Study
Arm/Group | Usual Care Comparison Condition - Children | Trauma-focused CBT Group Therapy - Children | Usual Care Comparison Condition - Caregivers | Trauma-focused CBT Group Therapy - Caregivers
Started | 320 | 320 | 320 | 320
Completed | 315 | 298 | 315 | 298
Not Completed | 5 | 22 | 5 | 22
Not completed — Lost to Follow-up | 5 | 1 | 5 | 1
Not completed — Withdrawal by Subject | 0 | 6 | 0 | 6
Not completed — Partial Intervention Completion | 0 | 15 | 0 | 15

BASELINE CHARACTERISTICS:
Population: Caregivers and Children were treated as dyads for the study, but have been categorized separately here for the purpose of reporting results.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care Comparison Condition - Children | Trauma-focused CBT Group Therapy - Children | Usual Care Comparison Condition - Caregivers | Trauma-focused CBT Group Therapy - Caregivers | Total
Number analyzed (Participants) | 320 | 320 | 320 | 320 | 1280
Age, Categorical [Count of Participants; unit: Participants] — Population: Child age missing for 2 comparison and 2 intervention participants.
  Participants
    number analyzed (Participants) | 318 | 318 | 320 | 320 | 1276
    <=18 years | 318 | 318 | 0 | 0 | 636
    Between 18 and 65 years | 0 | 0 | 298 | 292 | 590
    >=65 years | 0 | 0 | 22 | 28 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Child age missing for 2 comparison and 2 intervention participants.
  years
    number analyzed (Participants) | 318 | 318 | 320 | 320 | 1276
    (all) | 10.68 (1.66) | 10.58 (1.60) | 45.10 (13.34) | 44.43 (12.36) | 27.75 (19.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 160 | 160 | 288 | 286 | 894
  Male | 160 | 160 | 32 | 34 | 386
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 320 | 320 | 320 | 320 | 1280
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 320 | 320 | 320 | 320 | 1280
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Tanzania | 160 | 160 | 160 | 160 | 640
  Kenya | 160 | 160 | 160 | 160 | 640

OUTCOME MEASURES:

1. Primary Outcome: Posttraumatic Stress Syndrome (PTSS)
Description: Measured using the Child PTSD Symptoms Scale (CPSS). Caregiver and Child reported separately. Scale range 0-57, with 57 representing extremely high PTSS symptomatology (worse outcome). 634 children and 634 caregivers (1268 total) analyzed at baseline and 3-month follow-up--includes all 1280 enrolled at baseline, minus 12 lost to follow-up.
Time Frame: Baseline, 3 months
Population: Children and Caregivers from both comparison and intervention groups in all study settings (Tanzania and Kenya, rural and urban)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Tanzania Rural Comparison Child; Tanzania Urban Comparison Child; Kenya Rural Comparison Child; Kenya Urban Comparison Child; Tanzania Rural Comparison Caregiver; Tanzania Urban Comparison Caregiver; Kenya Rural Comparison Caregiver; Kenya Urban Comparison Caregiver: Half of the participating child/caregiver dyads will receive no intervention (usual care) to serve as a control.
- Tanzania Rural TF-CBT Child; Tanzania Urban TF-CBT Child; Kenya Rural TF-CBT Child; Kenya Urban TF-CBT Child; Tanzania Rural TF-CBT Caregiver; Tanzania Urban TF-CBT Caregiver; Kenya Rural TF-CBT Caregiver; Kenya Urban TF-CBT Caregiver: Half of the participating child/caregiver dyads will receive the 12-week Trauma-focused Cognitive Behavioral Therapy (TF-CBT) group treatment.
  Trauma-focused Cognitive Behavioral Therapy
Arm/Group | Tanzania Rural Comparison Child | Tanzania Urban Comparison Child | Tanzania Rural TF-CBT Child | Tanzania Urban TF-CBT Child | Kenya Rural Comparison Child | Kenya Urban Comparison Child | Kenya Rural TF-CBT Child | Kenya Urban TF-CBT Child | Tanzania Rural Comparison Caregiver | Tanzania Urban Comparison Caregiver | Tanzania Rural TF-CBT Caregiver | Tanzania Urban TF-CBT Caregiver | Kenya Rural Comparison Caregiver | Kenya Urban Comparison Caregiver | Kenya Rural TF-CBT Caregiver | Kenya Urban TF-CBT Caregiver
Number analyzed (Participants) | 64 | 91 | 63 | 96 | 64 | 96 | 64 | 96 | 64 | 91 | 63 | 96 | 64 | 96 | 64 | 96
score on a scale
  Baseline Score | 23.41 [21.61 to 25.21] | 21.23 [20.02 to 22.44] | 25.66 [23.99 to 27.32] | 23.40 [22.25 to 24.54] | 24.61 [22.74 to 26.47] | 22.03 [20.63 to 23.43] | 24.86 [22.91 to 26.81] | 24.70 [23.43 to 25.96] | 18.92 [17.13 to 20.72] | 18.81 [17.16 to 20.46] | 21.33 [19.35 to 23.31] | 22.08 [20.59 to 23.58] | 23.39 [21.11 to 25.67] | 20.61 [19.08 to 22.15] | 23.69 [22.07 to 25.30] | 21.98 [20.72 to 23.24]
  Post-Treatment Score | 8.98 [7.40 to 10.57] | 12.78 [11.17 to 14.39] | 10.17 [8.26 to 12.08] | 10.82 [9.26 to 12.38] | 22.44 [20.06 to 24.81] | 15.92 [14.57 to 17.26] | 14.00 [12.59 to 15.41] | 12.82 [11.52 to 14.12] | 6.94 [5.77 to 8.10] | 9.75 [8.43 to 11.07] | 5.56 [4.83 to 6.30] | 7.80 [6.69 to 8.91] | 23.06 [21.08 to 25.04] | 14.71 [13.29 to 16.13] | 10.77 [9.20 to 12.33] | 9.94 [8.90 to 10.97]
  Mean Change in Score | -14.40 [-16.55 to -12.24] | -8.39 [-10.19 to -6.60] | -15.48 [-17.43 to -13.54] | -12.53 [-14.17 to -10.88] | -2.17 [-5.14 to 0.80] | -6.11 [-7.76 to -4.47] | -10.86 [-13.40 to -8.32] | -11.88 [-13.41 to -10.34] | -11.81 [-13.63 to -9.98] | -8.77 [-10.56 to -6.98] | -15.77 [-17.78 to -13.75] | -14.23 [-16.07 to -12.39] | -0.33 [-3.24 to 2.58] | -5.91 [-7.78 to -4.03] | -12.92 [-15.19 to -10.65] | -12.04 [-13.48 to -10.61]

2. Primary Outcome: Childhood Traumatic Grief
Description: Measured using the Inventory of Complicated Grief (ICG). Child report only. Scale range 0-112, with 112 representing extremely high grief symptomatology (worse outcome). 634 children and 634 caregivers (1268 total) analyzed at baseline and 3-month follow-up--includes all 1280 enrolled at baseline, minus 12 lost to follow-up.
Time Frame: Baseline, 3 months
Population: Children from both comparison and intervention groups in all study settings (Tanzania and Kenya, rural and urban)
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Groups:
- Tanzania Rural Comparison Child; Tanzania Urban Comparison Child; Kenya Rural Comparison Child; Kenya Urban Comparison Child: Half of the participating children will receive no intervention (usual care) to serve as a control.
- Tanzania Rural TF-CBT Child; Tanzania Urban TF-CBT Child; Kenya Rural TF-CBT Child; Kenya Urban TF-CBT Child: Half of the participating children will receive the 12-week Trauma-focused Cognitive Behavioral Therapy (TF-CBT) group treatment.
  Trauma-focused Cognitive Behavioral Therapy
Arm/Group | Tanzania Rural Comparison Child | Tanzania Urban Comparison Child | Tanzania Rural TF-CBT Child | Tanzania Urban TF-CBT Child | Kenya Rural Comparison Child | Kenya Urban Comparison Child | Kenya Rural TF-CBT Child | Kenya Urban TF-CBT Child
Number analyzed (Participants) | 64 | 91 | 63 | 96 | 64 | 96 | 64 | 96
Score on a scale
  Baseline Score | 43.14 [38.18 to 48.10] | 40.63 [37.65 to 43.61] | 49.17 [43.98 to 54.37] | 44.73 [41.19 to 48.26] | 42.48 [37.70 to 47.27] | 38.34 [35.11 to 41.58] | 44.38 [38.98 to 49.77] | 42.46 [39.09 to 45.83]
  Post-Treatment Score | 13.44 [9.93 to 16.96] | 22.90 [19.09 to 26.72] | 16.00 [11.07 to 20.93] | 18.97 [15.75 to 22.18] | 38.13 [32.74 to 43.51] | 25.19 [22.13 to 28.25] | 21.09 [18.17 to 24.01] | 20.32 [17.25 to 23.39]
  Mean Change in Score | -29.65 [-35.42 to -23.88] | -17.25 [-20.97 to -13.54] | -33.17 [-38.20 to -28.15] | -25.77 [-29.98 to -21.55] | -4.36 [-11.12 to 2.40] | -13.01 [-17.15 to -8.88] | -23.28 [-29.76 to -16.80] | -22.14 [-26.06 to -18.21]

3. Secondary Outcome: Behavioral Difficulties
Description: Child report: Measured using the combined mean score of 1) the broadband externalizing scale of the Youth Self-Report (YSR) and 2) behavior-related items developed locally that are culturally specific. All items included are measured on a scale of 0-2, with 0 representing no behavioral difficulties (better) and 2 representing frequent behavioral difficulties (worse).
  Caregiver report: Measured using the combined mean score of 1) the broadband externalizing scale of the Child Behavior Checklist (CBCL) and 2) behavior-related items developed locally that are culturally specific. All items included are measured on a scale of 0-2, with 0 representing no behavioral difficulties (better) and 2 representing frequent behavioral difficulties (worse).
Time Frame: Baseline, 3 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Tanzania Rural Comparison Child | Tanzania Urban Comparison Child | Tanzania Rural TF-CBT Child | Tanzania Urban TF-CBT Child | Kenya Rural Comparison Child | Kenya Urban Comparison Child | Kenya Rural TF-CBT Child | Kenya Urban TF-CBT Child | Tanzania Rural Comparison Caregiver | Tanzania Urban Comparison Caregiver | Tanzania Rural TF-CBT Caregiver | Tanzania Urban TF-CBT Caregiver | Kenya Rural Comparison Caregiver | Kenya Urban Comparison Caregiver | Kenya Rural TF-CBT Caregiver | Kenya Urban TF-CBT Caregiver
Number analyzed (Participants) | 64 | 91 | 63 | 96 | 64 | 96 | 64 | 96 | 64 | 91 | 63 | 96 | 64 | 96 | 64 | 96
Score on a scale
  Baseline Score | 0.07 [0.05 to 0.09] | 0.11 [0.09 to 0.13] | 0.11 [0.08 to 0.14] | 0.11 [0.09 to 0.14] | 0.13 [0.09 to 0.16] | 0.15 [0.12 to 0.18] | 0.18 [0.13 to 0.23] | 0.21 [0.17 to 0.26] | 0.15 [0.12 to 0.17] | 0.16 [0.14 to 0.19] | 0.12 [0.10 to 0.15] | 0.17 [0.14 to 0.21] | 0.14 [0.10 to 0.17] | 0.18 [0.15 to 0.21] | 0.13 [0.09 to 0.16] | 0.25 [0.21 to 0.29]
  Post-Treatment Score | 0.06 [0.05 to 0.07] | 0.09 [0.07 to 0.10] | 0.08 [0.06 to 0.09] | 0.06 [0.05 to 0.08] | 0.13 [0.10 to 0.16] | 0.09 [0.07 to 0.12] | 0.11 [0.06 to 0.16] | 0.14 [0.10 to 0.18] | 0.12 [0.09 to 0.15] | 0.10 [0.08 to 0.12] | 0.09 [0.07 to 0.10] | 0.09 [0.07 to 0.10] | 0.16 [0.12 to 0.21] | 0.13 [0.11 to 0.16] | 0.11 [0.08 to 0.15] | 0.14 [0.12 to 0.17]
  Mean Change in Score | -0.01 [-0.03 to 0.01] | -0.02 [-0.04 to -0.00] | -0.03 [-0.07 to -0.00] | -0.05 [-0.08 to -0.02] | 0.00 [-0.04 to 0.05] | -0.05 [-0.09 to -0.02] | -0.07 [-0.12 to -0.01] | -0.07 [-0.13 to -0.01] | -0.03 [-0.06 to 0.01] | -0.07 [-0.09 to -0.04] | -0.02 [-0.06 to -0.01] | -0.09 [-0.12 to -0.05] | 0.03 [-0.02 to 0.07] | -0.05 [-0.08 to -0.02] | -0.02 [-0.05 to 0.02] | -0.11 [-0.15 to -0.08]

4. Other Pre Specified Outcome: Depression
Description: Child report: Measured using the combined mean score of 1) the broadband internalizing scale of the Youth Self-Report (YSR) and 2) depression-related items developed locally that are culturally specific. All items included are measured on a scale of 0-2, with 0 representing no depression (better) and 2 representing frequent signs of depression (worse).
  Caregiver report: Measured using the combined mean score of 1) the broadband internalizing scale of the Child Behavior Checklist (CBCL) and 2) depression-related items developed locally that are culturally specific. All items included are measured on a scale of 0-2, with 0 representing no depression (better) and 2 representing frequent signs of depression (worse).
Time Frame: Baseline, 3 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Tanzania Rural Comparison Child | Tanzania Urban Comparison Child | Tanzania Rural TF-CBT Child | Tanzania Urban TF-CBT Child | Kenya Rural Comparison Child | Kenya Urban Comparison Child | Kenya Rural TF-CBT Child | Kenya Urban TF-CBT Child | Tanzania Rural Comparison Caregiver | Tanzania Urban Comparison Caregiver | Tanzania Rural TF-CBT Caregiver | Tanzania Urban TF-CBT Caregiver | Kenya Rural Comparison Caregiver | Kenya Urban Comparison Caregiver | Kenya Rural TF-CBT Caregiver | Kenya Urban TF-CBT Caregiver
Number analyzed (Participants) | 64 | 91 | 63 | 96 | 64 | 96 | 64 | 96 | 64 | 91 | 63 | 96 | 64 | 96 | 64 | 96
Score on a scale
  Baseline Score | 0.23 [0.18 to 0.29] | 0.11 [0.09 to 0.13] | 0.41 [0.29 to 0.53] | 0.11 [0.09 to 0.14] | 0.52 [0.40 to 0.63] | 0.50 [0.43 to 0.57] | 0.63 [0.52 to 0.74] | 0.66 [0.57 to 0.74] | 0.21 [0.19 to 0.24] | 0.16 [0.14 to 0.19] | 0.20 [0.17 to 0.24] | 0.17 [0.14 to 0.21] | 0.48 [0.39 to 0.56] | 0.48 [0.42 to 0.54] | 0.48 [0.41 to 0.55] | 0.58 [0.52 to 0.64]
  Post-Treatment Score | 0.18 [0.15 to 0.22] | 0.09 [0.07 to 0.10] | 0.21 [0.17 to 0.25] | 0.06 [0.05 to 0.08] | 0.53 [0.40 to 0.63] | 0.38 [0.31 to 0.45] | 0.30 [0.22 to 0.38] | 0.33 [0.27 to 0.39] | 0.17 [0.15 to 0.19] | 0.10 [0.08 to 0.12] | 0.15 [0.13 to 0.17] | 0.09 [0.07 to 0.10] | 0.55 [0.48 to 0.62] | 0.36 [0.30 to 0.41] | 0.28 [0.24 to 0.32] | 0.32 [0.28 to 0.36]
  Mean Change in Score | -0.05 [-0.11 to 0.01] | -0.02 [-0.04 to -0.00] | -0.21 [-0.32 to -0.10] | -0.05 [-0.08 to -0.02] | 0.01 [-0.16 to 0.18] | -0.11 [-0.20 to -0.03] | -0.33 [-0.48 to -0.19] | -0.32 [-0.43 to -0.22] | -0.04 [-0.08 to -0.01] | -0.07 [-0.09 to -0.04] | -0.05 [-0.09 to -0.02] | -0.09 [-0.12 to -0.05] | 0.07 [-0.03 to 0.18] | -0.12 [-0.19 to -0.05] | -0.20 [-0.28 to -0.13] | -0.26 [-0.33 to -0.19]

5. Other Pre Specified Outcome: Child Functioning
Description: Locally developed tool used to measure functional impairment and improvement over time.
Time Frame: Baseline, 3 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Child-Guardian Relationship
Description: Measured using the Child-Parent Relationship Scale (CPRS)
Time Frame: Baseline, 3 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year, 3 months
Groups:
- Trauma-focused CBT Group Therapy: Half of the participating children/guardian dyads will receive the 12-week Trauma-focused Cognitive Behavioral Therapy (TF-CBT) group treatment.
  Trauma-focused Cognitive Behavioral Therapy
Arm/Group | Usual Care Comparison Condition | Trauma-focused CBT Group Therapy
All-Cause Mortality (participants affected / at risk) | 0/640 | 0/640
Serious Adverse Events (participants affected / at risk) | 0/640 | 0/640
Other Adverse Events (participants affected / at risk) | 0/640 | 0/640

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-05-03): https://cdn.clinicaltrials.gov/large-docs/66/NCT01822366/Prot_SAP_000.pdf